CLINICAL TRIAL: NCT02123875
Title: Family-led Rehabilitation After Stroke in India
Brief Title: ATTEND-Family-led Rehabilitation After Stroke in India
Acronym: ATTEND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christian Medical College and Hospital, Ludhiana, India (Other)
Collaborators: The George Institute for Global Health, Australia (Other)
Responsible Party: Principal Investigator, jeyarajpandian, Professor and Head, Department of Neurology, Christian Medical College and Hospital, Ludhiana, India
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0001
Record Dates: First submitted 2014-04-11; First posted 2014-04-28 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control arm (Other): Routine hospital based physiotherapy
  Interventions: Other: Control arm
- Physiotherapy intervention arm (Other): Caregiver delivered, home based physiotherapy
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy
  Arms: Physiotherapy intervention arm
Other: Control arm — Routine hospital based physiotherapy
  Arms: Control arm

SUMMARY:
ATTEND Trial is based on early supported discharge- home based stroke rehabilitation model which proves to offer several advantages in low and mid income countries. The objectives of the pilot stude were to determine that with a randomized blinded outcome assessor, controlled trial, family- led caregiver- delivered home based rehabilitation is better than usual care for those with disabling stroke in India and the feasibility of this model.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years)
* Recent (<1 month) acute ischaemic/haemorrhagic/ undifferentiated stroke
* Residual disability (requiring help from another person for everyday activities)
* Expected to survive to discharge from hospital with a reasonable expectation of six month survival
* Able (or by proxy) to provide informed consent

Exclusion Criteria:

* Unable to identify a suitable family - nominated caregiver for training and subsequent delivery of care
* Those unwilling/unable to adhere to follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2011-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change in modified Rankin Score | 3rd and 6th month

CONTACTS AND LOCATIONS:
Overall Officials: Jeyaraj D Pandian, MD DM FRACP, Principal Investigator — Christian Medical College and Hospital
Locations (1):
- Christian Medical College and Hospital, Ludhiana, Punjab, India

REFERENCES:
- [Derived] Crocker TF, Brown L, Lam N, Wray F, Knapp P, Forster A. Information provision for stroke survivors and their carers. Cochrane Database Syst Rev. 2021 Nov 23;11(11):CD001919. doi: 10.1002/14651858.CD001919.pub4. PMID 34813082
- [Derived] Wang X, Moullaali TJ, Li Q, Berge E, Robinson TG, Lindley R, Zheng D, Delcourt C, Arima H, Song L, Chen X, Yang J, Chalmers J, Anderson CS, Sandset EC. Utility-Weighted Modified Rankin Scale Scores for the Assessment of Stroke Outcome: Pooled Analysis of 20 000+ Patients. Stroke. 2020 Aug;51(8):2411-2417. doi: 10.1161/STROKEAHA.119.028523. Epub 2020 Jul 9. PMID 32640944